CLINICAL TRIAL: NCT04939545
Title: Efficacy of Surgically Placed Intercostal Catheter (ICC) for Postoperative Analgesia After Minimally Invasive Anatomical Lung Resection Using Ropivacaine: A Randomised, Double-blind, Placebocontrolled, Superiority Study
Brief Title: Study of Postoperative ICC Analgesia
Acronym: SPICA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-00922; kt21Lardinois
Record Dates: First submitted 2021-06-09; First posted 2021-06-25 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Analgesia
Keywords: Surgically Placed Intercostal Catheter (ICC); minimally invasive anatomical lung resection; ropivacaine; loco-regional analgesia; thoracic analgesia; Video-assisted thoracoscopic surgery (VATS)
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective, placebo-controlled, randomised, double-blind, superiority
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators, care providers, data analyst and trial participants are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention Ropivacain (Experimental): Ropivacain Fresenius 0.2% is a solution for infusion/ injection and will be continuously administered with an elastomer pump through the surgically placed intercostal catheter (ICC) between parietal pleura and fascia endo-thoracica at the level of surgical incision for a maximum of 72 hours at an initial standard flow rate setting of 6 ml/h using 2 mg/ml ropivacaine. In case pain exceeds 7 on NRS later than 2 hours after skin closure the flow rate will be adjusted on 8 ml/h. Furthermore, Ropivacain Fresenius 0.2% will be provided in a 20 ml glass vial for flushing the infusion line and subpleural administration.
  Interventions: Drug: Ropivacain
- Control Intervention Placebo (Placebo Comparator): Placebo (NaCl 0.9% B. Braun) is an isotonic solution for infusion and will be continuously administered with an elastomer pump through the surgically placed intercostal catheter (ICC) between parietal pleura and fascia endo-thoracica at the level of surgical incision for a maximum of 72 hours at an initial standard flow rate setting of 6 ml/h using NaCl 0.9%. In case pain exceeds 7 on NRS later than 2 hours after skin closure the flow rate will be adjusted on 8 ml/h. Furthermore, NaCl 0.9% will be provided in a 20 ml glass vial for flushing the infusion line and for subpleural administration, which will be prepared by the hospital pharmacy.
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Ropivacain — Intercostal continuous loco-regional ropivacaine (2 mg/ml) administration over an elastomeric pump through a surgically placed intercostal catheter (ICC) for a maximum of 72h.
  As concomitant treatments a standardized anesthesia protocol including intravenous continuous application of propofol and remifentanil is used. Additionally, i.v. metamizol at a dose of 1 g will be administered at the end of surgery as a standard, if not contraindicated.
  In a standardized postoperative pain protocol the use of basic oral medication is documented as part of the postoperative follow-up and consists of:
  ibuprofen 3 x 400 mg p. o. for 3 days, metamizol 4 x 1 g p. o. for 3 days; if ibuprofen and/or metamizol contraindicated then paracetamol p. o. 3 x 1g for 3 days will be administered; morphine 10 mg p. o. 6 times daily will be given on a patient demand basis.
  Arms: Experimental Intervention Ropivacain
Drug: NaCl 0.9% — Intercostal continuous loco-regional placebo solution (NaCl 0,9%) administration over an elastomeric pump through a surgically placed intercostal catheter (ICC) for a maximum of 72h. As concomitant treatments a standardized anesthesia protocol including intravenous continuous application of propofol and remifentanil is used. Additionally, i.v. metamizol at a dose of 1 g will be administered at the end of surgery as a standard, if not contraindicated.
  In a standardized postoperative pain protocol the use of basic oral medication is documented as part of the postoperative follow-up and consists of:
  ibuprofen 3 x 400 mg p. o. for 3 days, metamizol 4 x 1 g p. o. for 3 days; if ibuprofen and/or metamizol contraindicated then paracetamol p. o. 3 x 1g for 3 days will be administered; morphine 10 mg p. o. 6 times daily will be given on a patient demand basis.
  Arms: Control Intervention Placebo

SUMMARY:
This study is to examine the analgesic effectiveness of continuous loco-regional analgesic application (ropivacaine) through surgically placed Intercostal Catheter (ICC) and to establish correctly this method as a possible standard of care in the postoperative analgesia after Video-assisted thoracoscopic surgery (VATS) anatomical lung resection.

DETAILED DESCRIPTION:
Good control of the pain without excessive use of opiates supports the benefits of minimally invasive surgical procedure.

This study is to examine the efficacy of continuously via surgically placed intercostal catheter administered ropivacaine at a flow rate of 6-8 ml/h of 2 mg/ml on post-operative pain (NRS) and pulmonary function (FEV1, PEF) during a maximum of 72 ± 2 hours after skin closure. Patients undergoing video-assisted thoracoscopic anatomical resection of the lung under general anaesthesia with confirmed or anticipated Stage I Lung cancer will be included. The study will be conducted as superiority, double-blind, placebo-controlled, randomized. The efficacy of loco-regional administered ropivacaine will be compared to placebo (NaCl, 0.9%) administration. The whole study period per participant is expected to be 6 months. In the follow-up, 6 months after surgery, the impact of ropivacaine on long-term pain (NRS, McGill) and pulmonary function (FEV1, PEF) shall be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Patient undergoing video-assisted thoracoscopic anatomical resection of the lung under general anaesthesia for confirmed or anticipated Stage I lung cancer (UICC 8th edition)
* American Society of Anesthesiologists (ASA) physical status classes I to III

Exclusion Criteria:

* NRS while coughing > 0
* Previous ipsilateral thoracotomy or sternotomy
* Abdominal or contralateral thoracic surgery up to 6 months preoperatively
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product
* Contraindications to self-administration of opioids
* Women who are pregnant or breast feeding
* Chronic steroid therapy (e.g. Prednisone > 10mg/day for more than last 2 weeks before surgery)
* Chronic, daily pain therapy
* Congestive heart failure
* Liver insufficiency
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Enrolment of the investigator, his/her family members, employees and other dependent person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
change in pain numerical rating scale (NRS) while coughing | before surgery, at 2, 4, 8, 24, 48, 72 hours after skin closure
  change in pain NRS (scale 0-10) while coughing in the Ropivacaine arm compared to Placebo arm; 0 = no pain to 10 = worst pain imaginable

SECONDARY OUTCOMES:
change in pain NRS at rest | before surgery, at 2, 4, 8, 24, 48 and 72 hours after skin closure, 1 day before hospital discharge and 6 months ± 28 days after surgery
  change in pain NRS at rest in the Ropivacaine arm compared to Placebo arm; 0 = no pain to 10 = worst pain imaginable
number of daily postoperative pain killer consumption | within 72 ± 2 hours postoperative
  number of daily postoperative pain killer consumption
change in Silverman integrating approach (SIA) score, combined rank-based analysis of pain score and opioid consumption. | within 72 ± 2 hours postoperative
  Silverman integrating approach (SIA) score is a combined score from the pain numerical rating scale (NRS) and analgesics (opiate) usage. It is a sum of rank- based percentage differences from the mean rank in pain scores and opioid use, ranging from -200 to 200%. SIA-scores integrate pain scores and opioid use for the individual patient.
change in forced expiratory volume in 1 second (FEV1) | before surgery, at 24, 48 and 72 hours after skin closure, 1 day before hospital discharge and 6 months ± 28 days after surgery
  change in forced expiratory volume in 1 second (FEV1)
change in peek expiratory flow (PEF) | before surgery, at 24, 48 and 72 hours after skin closure, 1 day before hospital discharge and 6 months ± 28 days after surgery
  change in peek expiratory flow (PEF)
change in the short-form McGill Questionnaire (SF-MPQ) | before surgery, 48 hours after skin closure and 6 months ± 28 days after surgery
  The SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors. The SF-MPQ also includes the Present Pain Intensity (PPI) index of the standard MPQ and a 10 cm visual analogue scale (VAS), 0 = no pain to 10 = worst pain imaginable. The higher the integrated score, the higher the pain level.
Patient Controlled Analgesia (PCA) demand | within 72 ± 2 hours postoperative
  PCA demand (Consumption of intravenous opiate)
duration of chest tube chest tube | within 72 ± 2 hours postoperative
  duration of chest tube
length of hospital stay | in the average within 30 days postoperative
  number of days in hospital postoperative
30 day mortality | within 30 days postoperative
  30 day mortality
number of gastrointestinal tract events | within 72 ± 2 hours postoperative
  postoperative nausea and vomiting
time to first defecation | in the average within 30 days postoperative
  time to first defecation

CONTACTS AND LOCATIONS:
Overall Officials: Didier Lardinois, Prof. Dr. med., Study Chair — University Hospital Basel, Division of Thoracic Surgery; Aljaz Hojski, Dr. med., Principal Investigator — University Hospital Basel, Division of Thoracic Surgery
Locations (1):
- University Hospital Basel, Department of Thoracic Surgery, Basel, Switzerland

REFERENCES:
- [Derived] Hojski A, Kramer M, Gecas P, Djakovic Z, Tsvetkov N, Mallaev M, Bolliger D, Lampart A, Lardinois D. The efficacy of loco-regional ropivacaine analgesia via intercostal catheters after lung resection: a randomized, double-blind, placebo-controlled, superiority study. Eur J Cardiothorac Surg. 2024 Oct 1;66(4):ezae342. doi: 10.1093/ejcts/ezae342. PMID 39352775